CLINICAL TRIAL: NCT00915629
Title: Prevention of Recurrent Vulvovaginal Candidiasis With Lactibiane Candisis 5M®
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2008-A01513-52
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Vaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotic (Experimental): Dietary supplement
  Interventions: Dietary Supplement: Lactibiane candisis 5M

INTERVENTIONS:
Dietary Supplement: Lactibiane candisis 5M — 2 gelules per day for 2 months then 1 gelule per day for 4 months

SUMMARY:
Vulvovaginal candidiasis (VVC) is a common infection among women that is associated with considerable morbidity and health-care cost. 75% of women will suffer of Candida infection for at least one time in their life. 20% of women who suffer from VVC will have ≥ 4 episodes of VVC during the one year prior to the survey. 80% of these VVC are caused by Candida albicans. Current treatments, based on imidazoles, face many failures or recurrences. The type of probiotic Lactobacillus may participate in the prevention of recurrent vulvo-vaginitis in reducing the proliferation of intestinal Candida albicans, its adherence to the vaginal walls, the potentiation of its propagation. The primary objective of this study was to investigate if our supplementary treatment could improve the initial cure rate after vaginal econazole therapy.

ELIGIBILITY:
Inclusion Criteria:

* women
* 18-65 years
* suffering from 4 or more episodes of VVC during the 1 year prior to the survey
* all participants must be symptomatic with a microbiological proof of infection with candida albicans

Exclusion Criteria:

* Pregnancy, lactation being
* HIV infection, chemotherapy or illness serious enough to induce an immune deficiency. A diabetic patient will not be systematically excluded;
* Vulvo-vaginitis and / or cervicitis specific, defined in a bacteriological examination by the presence of herpes virus, gonorrhea or chlamydia;
* Bacterial Vaginosis or Trichomonas;
* Use of vaginal probiotics in the months before inclusion;
* Cure of probiotics in the months preceding the inclusion;
* Contraindication to Gynopévaryl LP

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to investigate if Lactibiane candisis 5M supplementation could lengthen the time to relapse after initial local cure | 9 months

SECONDARY OUTCOMES:
The secondary objective of this study is to compare the number of recurrence in the lactibiane candisis 5M group versus placebo. | 2, 3, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: AZOULAY Catherine, MD, Principal Investigator
Locations (1):
- Pileje, Paris, France

REFERENCES:
- [Derived] Cooke G, Watson C, Deckx L, Pirotta M, Smith J, van Driel ML. Treatment for recurrent vulvovaginal candidiasis (thrush). Cochrane Database Syst Rev. 2022 Jan 10;1(1):CD009151. doi: 10.1002/14651858.CD009151.pub2. PMID 35005777